CLINICAL TRIAL: NCT06515652
Title: To Compre the Efficacy and Safety of Herbal Medicine With Allopathic Therapy for Metabolic Syndrome: A Randomized , Multi-center, Clinical Study
Brief Title: To Compare the Effects of Herbal Medicines With Traditional Allopathic Medicines in Cases of Patients With Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, SYEDA AMBER ZAIDI, Assitstant Professor, Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHMS HamdardUniversity
Record Dates: First submitted 2024-07-02; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome
Keywords: Hyperlipidemia; Type 2 Diabetes; Hypertension; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Hyperlipidemias; Diabetes Mellitus, Type 2; Hypertension; Obesity | interventions — Rosuvastatin Calcium; Metformin; Sitagliptin Phosphate; Telmisartan; ginger extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allopathic (Active Comparator): 1. Tablet.Rosuvastatin 10mg once daily for 3 months
  2. Tablet. Telmisartan 40mg once daily for 3 months
  3. Tablet. Sitagliptin / Metformin 50/500mg once daily for 3 months
  Interventions: Drug: rosuvastatin, METFORMIN, Sitagliptin, Telmisartan, Cinnamon. garlic, Ginger, Methi dana, Arjun
- Herbal (Active Comparator): 1. Cinammon powder 2 gm once daily for 3 months
  2. Garlic powder 1 gm once daily for 3 months
  3. Ginger powder 4 gm once daily for 3 months
  4. Fenugreek powder 10 gm once daily for 3 months
  5. Arjuna 2 gm once daily for 3 months
  Interventions: Drug: rosuvastatin, METFORMIN, Sitagliptin, Telmisartan, Cinnamon. garlic, Ginger, Methi dana, Arjun

INTERVENTIONS:
Drug: rosuvastatin, METFORMIN, Sitagliptin, Telmisartan, Cinnamon. garlic, Ginger, Methi dana, Arjun — Comparing allopathic and herbal group of drugs for metabolic syndrome

SUMMARY:
Metabolic syndrome is an important global public health problem and comprises a group of complex risk factors, including obesity, dyslipidemia, hyperglycemia, and hypertension. One of the main diagnostic components of metabolic syndrome is obesity, which is usually measured by the waist circumference and the intra-abdominal visceral fat, in addition to dyslipidemia (the condition of raised triglycerides and reduced high density lipoprotein (HDL)-cholesterol in blood; other components are raised blood pressure and fasting plasma glucose, all of which are related to weight gain.

Metabolic syndrome is related to cardio metabolic risk factors and lipid disorders. Worldwide, cardiovascular diseases (CVD) are the leading cause of mortality and morbidity. It is expected that by 2030, mortality from CVD will reach 22.5 million people, compared with 17.5 million deaths in 2012.

Major pharmacological interventions include management of dyslipidemia with statins, decreasing prothrombotic risk with antiplatelet drugs, and the use of insulin sensitizers to decrease the risk of diabetes. In addition to non-pharmacologic interventions that improve BP, pharmacological agents provide the primary basis for hypertension management in the majority of patients. Among major antihypertensive agents, angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), calcium channel blockers (CCBs), and thiazide (or thiazide-like) diuretics are preferentially recommended in the general condition because of their additional cardiovascular protection effects and/or accessibility.

Herbal drugs are being used worldwide in the management of metabolic syndrome now a days. Some of the herbs e.g. Terminalia arjuna, Trigonella Foenum-graecum, Allium Sativum, Cinnamon verum and Zingiber Officinale are being used very effectively in managing metabolic syndrome.

METHODOLOGY:

The basic purpose of this study will be to explore a poly herbal combination for effective and safe management of metabolic syndrome. This is a multicenter; prospective study will be conducted in the department of Pharmacology, HCMD in collaboration with Hamdard University Hospital, National Medical Center and Amna Unani Hospital.

After fulfilling the inclusion and exclusion criteria a total of 200 patients will be enrolled and divided in 2 groups. One group will be given allopathic combination while the other group will be given a poly herbal formulation. Important parameters include BMI, Systolic and Diastolic blood pressure, lipid profile, HbA1c, S.creatinine, Urinary Albumin, Urinary Creatinine, ALT & AST. Follow up will be done at day 0, 30, 60 & 90th of treatment. The data will be recorded in a tabulated form and statistical analysis will be done at the end of the study to see the significance of the two studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients ageing between 35-65 years;
* Patients with a diagnosis of metabolic syndrome according to the criteria of IDF 2005

Exclusion Criteria:

* Pregnant & lactating female
* Use of insulin or sulfonamide derivative oral antidiabetic drugs
* Doing heavy physical activity or working in a physically demanding job
* Presence of liver or kidney disease, or immune deficiency
* Patients with history of myocardial infarction, coronary artery bypass surgery, unstable angina & cardiac failure.
* Conditions that will seriously affect weight management such as having had bariatric surgery
* Determined to have had an unintentional sudden weight loss of more than 5% in the last three months
* Intellectual disability or significant medical or psychiatric illness as documented by the referring doctor.
* Any contraindication to the use of drugs involved in the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin | 3 months
  at day 0 and day 90
Systolic blood pressure, diastolic blood pressure | 3 months
  at day 0, day 30, day 60 and day 90
triglyceride level | 3 months
  at day 0, day 30, day 60 and day 90
high density lipoprotein level | 3 months
  at day 0, day 30, day 60 and day 90
waist hip ratio | 3 months
  at day 0 and day 90

SECONDARY OUTCOMES:
Fasting blood sugar, random blood sugar | 3 months
  at day 0, day 30, day 60 and day 90
serum cholesterol level | 3 months
  at day 0, day 30, day 60 and day 90
serum creatinine level | 3 months
  at day 0, day 30, day 60 and day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. M. Sajid Abbas Jaffri, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No